CLINICAL TRIAL: NCT01116089
Title: PHARMACOKINETIC STUDY OF BRAMITOB® ADMINISTERED FOR INHALATION BY PARI eFLOW® RAPID ELECTRONIC NEBULIZER VS PARI LC® PLUS NEBULIZER COUPLED WITH THE PARI TURBO BOY® N COMPRESSOR IN CYSTIC FIBROSIS PATIENTS INFECTED WITH PSEUDOMONAS AERUGINOSA
Brief Title: Pharmacokinetic Study of Bramitob® Administered for Inhalation by PARI eFlow® vs PARI LC® PLUS Nebulizer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-0908-PR-0029; 2009-016780-11 (EudraCT Number)
Record Dates: First submitted 2010-04-29; First posted 2010-05-04 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis, tobramycin,nebulizer, PK
MeSH Terms: conditions — Cystic Fibrosis | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PARI LC® PLUS nebulizer (Active Comparator)
  Interventions: Drug: Bramitob® administered by PARI LC® PLUS nebulizer
- PARI eFlow® rapid electronic nebulizer (Active Comparator)
  Interventions: Drug: Bramitob® administered by PARI eFlow® rapid electronic nebulizer

INTERVENTIONS:
Drug: Bramitob® administered by PARI LC® PLUS nebulizer — (tobramycin 300mg /4mL) solution administered by inhalation twice daily for 28 days
  Other Names: Bramitob®, Tobrineb®, Actitob®
  Arms: PARI LC® PLUS nebulizer
Drug: Bramitob® administered by PARI eFlow® rapid electronic nebulizer — (tobramycin 300mg /4mL) solution administered by inhalation twice daily for 28 days
  Other Names: Bramitob®, Tobrineb®,Actitob®
  Arms: PARI eFlow® rapid electronic nebulizer

SUMMARY:
The purpose of this study is to assess pharmacokinetic and safety comparability of Bramitob® when administered for inhalation by using PARI eFlow® rapid electronic nebulizer vs PARI LC® PLUS nebulizer in Cystic Fibrosis Patients infected with Pseudomonas Aeruginosa

ELIGIBILITY:
Main inclusion Criteria:

* Patients of either sex aged ≥ 18 years;
* Clinical diagnosis of cystic fibrosis (patients registered in the National Registry of cystic fibrosis or other documents, if applicable, depending on country legislation);
* Positive response (sweat chloride concentration ≥ 60 mmol/l) in the standard sweat test documented in the clinical records or sweat chloride concentration ≥ 40 mmol/l and at least two gene mutations consistent with CF documented in the clinical records;
* Chronic colonization of Pseudomonas aeruginosa
* FEV1 ≥ 35% of the predicted normal value calculated according to the recommendation of the Official Statement of the European Respiratory Society and American Thoracic Society

Main exclusion Criteria:

* Evidence of impaired renal function (serum creatinine level ≥ 1.5 mg/dl);
* Evidence of impaired auditory function (auditory threshold in either ear above 20 dB at frequencies between 250 and 8000Hz);
* Sputum culture containing Burkholderia cepacia;
* Received loop diuretics within 7 days before study drug administration;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Plasma tobramycin pharmacokinetic parameters (Cmax and AUC0-t) after twice daily inhalation of Bramitob® using PARI eFlow® nebulizer vs PARI LC® PLUS nebulizer | on day 28

SECONDARY OUTCOMES:
Plasma tobramycin pharmacokinetic parameters (Cmax, tmax and AUC0-t) after inhalation of Bramitob® using PARI eFlow® nebulizer vs PARI LC® PLUS nebulizer | on day 1
Sputum tobramycin pharmacokinetic parameters (Cmax, tmax and AUC0-t) after inhalation of Bramitob® using PARI eFlow® nebulizer vs PARI LC® PLUS nebulizer | on day 1 and on day 28
Accumulation of tobramycin in plasma and sputum after repeated doses calculated as the ratio: AUC0-t DAY 28 / AUC0-t DAY 1 and Cmax DAY 28 / Cmax DAY 1 | day 1 - day 28
Safety assessed by adverse events, adverse drug reactions, incidence of bronchospasm, laboratory parameters, physical examination, body weight, vital signs results | day1-day28
Number of patients with minimum plasma tobramycin levels Cmin > 2mcg/mL and maximum plasma tobramycin levels Cmax > 12 mcg/mL | on day 28
Time necessary for the nebulization of the dose | on day 1 and on day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Ružička, MD, PhD, Principal Investigator — Fakultná nemocnica s poliklinikou Bratislava, Slovakia; Andrej Somos, MD, Principal Investigator — University Hospital of L. Pasteur, Pneumonology Department, Rastislavova 43, 041 90, Kosice, Slovakia; Jana Skřičková, MD, PhD, Principal Investigator — University Hospital Brno Bohunice, Jihlavská 20, 625 00, Brno, Czech Republic; Eva Beresova, M.D, Principal Investigator — University hospital with Health Center, F.D. Roosevelta Banská Bystrica, L. Svoboda´s square 1, 975 17, Banská Bystrica, Slovakia; Svetlana Şciuca, M.D, PhD, Principal Investigator — SMSI Institude of Cardiology, MD-2025, 29/1 Testimitanu str., Chisinau, Republic of Moldova
Locations (5):
- University Hospital Brno Bohunice, Brno, Czechia
- SMSI Institude of Cardiology, Chisinau, Moldova
- Slovakia (3):
  - University hospital with Health Center, Banská Bystrica
  - Fakultná nemocnica s poliklinikou Bratislava (FNsP), Brastislava
  - University Hospital of L. Pasteur, Pneumonology Department, Košice

REFERENCES:
- [Result] Govoni M, Poli G, Acerbi D, Santoro D, Cicirello H, Annoni O, Ruzicka J. Pharmacokinetic and tolerability profiles of tobramycin nebuliser solution 300 mg/4 ml administered by PARI eFlow((R)) rapid and PARI LC Plus((R)) nebulisers in cystic fibrosis patients. Pulm Pharmacol Ther. 2013 Apr;26(2):249-55. doi: 10.1016/j.pupt.2012.12.002. Epub 2012 Dec 8. PMID 23232039